CLINICAL TRIAL: NCT04737928
Title: Prospective, Single Center Switching Study of 0.0015% Tafluprost Ophthalmic Solution in Primary Open-angle Glaucoma and Ocular Hypertension Patients With Corneal Disorders
Brief Title: Prospective, Single Center Switching Study of 0.0015% Tafluprost Ophthalmic Solution in Primary Open-angle Glaucoma and Ocular Hypertension Patients With Corneal Disorders (Switching From 0.005% Latanoprost Ophthalmic Solution)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santen Pharmaceutical (Taiwan) Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TFT-IIR_TW001
Record Dates: First submitted 2021-01-28; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Glaucoma, Primary Open Angle
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Latanoprost; tafluprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- latanoprost switch to tafluprost (Experimental): POAG and OH patients prescribed latanoprost(QID) at least 3 months (IOP>20). At least one eye must have a score above 1 on the NEI scale. Switch to latanoprost (QID) for 3 months.
  Interventions: Drug: Latanoprost; Drug: tafluprost

INTERVENTIONS:
Drug: Latanoprost — latanoprost 0.05%(one drop, once daily)
Drug: tafluprost — tafluprost 0.015% (one drop, once daily)

SUMMARY:
The objective of this study was to investigate the improving effect of corneal disorder in primary open-angle glaucoma and ocular hypertension patients, when switched from the 0.005% latanoprost ophthalmic solution (one drop at a time, once daily) to the 0.0015% tafluprost ophthalmic solution (one drop at a time, once daily). Efficacy also was investigated.

ELIGIBILITY:
Inclusion Criteria:

* Age of 20 years or older and those who was provided informed consent.
* POAG or OH patients whose IOP did not exceed 22 mmHg at Visit 0.
* Patients had treated with prostaglandin ophthalmic solution (0.005% Latanoprost) for at least 3 months before enrollment.
* Patients who had corneal disorders due to the PG usage. (At least one eye had a score above 1 on the NEI scale)
* If only one eye was eligible, it was evaluated. When both eyes were eligible, then the eye with a higher NEI score was selected for evaluation.
* Outpatients who visited the clinic on the designated day as instructed by the physician.

Exclusion Criteria:

* Those with severe visual field disorder (Mean deviation of 15 dB or worse).
* Those who received corneal refractive surgery.
* Those with a history of ocular surgeries (such as corneal refractive surgery, intraocular surgery including ocular laser treatment which affected the patient's ocular surface condition) within 3 months prior to enrollment.
* Any corneal abnormality or other condition preventing IOP measurement.
* Those who used artificial tears to relieve dry eye symptoms.
* Those with severe dry eye, ocular allergy, ocular infection or ocular inflammation which considered affect interpretation of the results of the study. Those who used systemic or ophthalmic steroids (excluding topical skin steroidal ointment) and anti-glaucoma agents other than prostaglandin ophthalmic solution.
* Female patients who were pregnant, nursing or lactating.
* Those with a history of drug allergy (hypersensitivity) to the drugs to be used during the study period (anesthetic ophthalmic solution, fluorescein, etc.) or similar drugs to the study medication.
* Those who wore contact lenses during the study period.
* Those who had participation in another clinical trial involving an investigational drug/device, or participation in such a trial within the last 30 days.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Efficacy: Changes in the Intraocular Pressure (IOP) at each visit | 3 months
  Tonometer
Safety:Changes in the fluorescein staining score (NEI) at Visit 2 | 3 months
  fluorescein staining

SECONDARY OUTCOMES:
Changes in the fluorescein staining score (NEI) at Visit 1 | 1 months
  fluorescein staining
Changes in ocular symptoms (irritation/burning/stinging, foreign body sensation, tearing, itching and dry eye sensation) at each visit | 3 months
  Questionnaire
Changes in the Tear Break-Up Time (TBUT) at each visit | 3 months
  slit-lamp
Changes in the hyperaemia at each visit | 3 months
  slit-lamp
Treatment compliance | 3 months
  Questionnaire
Concomitant medication | 3 months
  Questionnaire
Patient satisfaction about test medication | 3 months
  Questionnaire
Usability of eyedrop bottle | 3 months
  Questionnaire
Adverse drug reactions | 3 months
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Chi Mei Hospital Liouying Branch, Tainan, Taiwan